CLINICAL TRIAL: NCT03788265
Title: Efficacy of Autologous Micro-fragmented Adipose Tissue Intra-articular Injection for Knee Osteoarthritis
Brief Title: Autologous Micro-fragmented Adipose Tissue Injection for Knee Osteoarthritis
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Second Affiliated Hospital, School of Medicine, Zhejiang University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: lipo-knee OA-dxs
Record Dates: First submitted 2018-11-14; First posted 2018-12-27 (Actual); Last update posted 2019-04-16 (Actual); Status verified 2019-04

CONDITIONS: Knee Osteoarthritis
MeSH Terms: conditions — Osteoarthritis, Knee

ARMS (1):
- injection (Experimental)
  Interventions: Device: Lipogems

INTERVENTIONS:
Device: Lipogems — harvest and inject micro-fragment adipose tissue

SUMMARY:
Knee osteoarthritis (OA) is characterized by loss of cartilage leading to instability, reduced range of motion, and functional limitations. Current treatment has various limitations so that alternative options to restore function and alleviate joint pain, with the ultimate goal of healing damaged articular cartilage are needed. Mesenchymal stem cells (MSCs) therapy has shown promising results. However, MSCs are limited by complex regulatory issues. Lipogems is a technique to harvest, process, and inject minimally manipulated adipose tissue through mild mechanical force. This procedure is enzyme free and requires no clonal expansion or manipulation. The goal of this study is to evaluate the possible benefits of reduced joint pain and increased joint functionality in patients with knee osteoarthritis after the injection of Lipogems.

ELIGIBILITY:
Inclusion Criteria:

* Age of eighteen or older
* Diagnosis of symptomatic knee osteoarthritis
* Radiographic evidence of knee osteoarthritis
* Failure of conservative treatment

Exclusion Criteria:

* Treatment with any intra-articular knee injection within 8 weeks before surgery
* Any disease or condition potential to interfere study outcome
* Under 18 years of age

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2016-01-01 (Actual); Primary Completion 2020-01-01 (Estimated); Study Completion 2021-01-01 (Estimated)

PRIMARY OUTCOMES:
Change in Visual Analog Pain Scale (VAS) Over Time | Pre-op, then post-op: 1 month, 3 months, 6 months, 1 year, 2 years
  Scaled pain score to assess change in a patient's knee pain over time. Pain level is marked on a 100 mm line with the 0 mm corresponding to "no pain" and the 100 mm corresponding to 10/10 pain. Using a ruler, the score is determined by measuring the distance (mm) on the 100 mm line between the "no pain" anchor and the patient's mark, providing a range of scores from 0-100. The following cut points on the pain VAS have been recommended: no pain (0-4 mm), mild pain(5-44 mm), moderate pain (45-74 mm), and severe pain (75-100 mm).

SECONDARY OUTCOMES:
Change in the knee injury and osteoarthritis score (KOOS) Over Time | Pre-op, then post-op: 1 month, 3 months, 6 months, 1 year, 2 years
  Patient self-reported outcome measure to assess the patient's opinion about their knee and associated issues. KOOS consists of 5 subscales; Pain, other Symptoms, Function in daily living (ADL), Function in sport and recreation (Sport/Rec) and knee related Quality of life (QOL). Standardized answer options are given (5 Likert boxes) and each question gets a score from 0 to 4. A normalized score (100 indicating no symptoms and 0 indicating extreme symptoms) is calculated by adding the subscales together.

CONTACTS AND LOCATIONS:
Locations (1):
- Second affiliated hospital, school of medicine, Zhejiang Uni., Hangzhou, Zhejiang, China